CLINICAL TRIAL: NCT01264445
Title: A Phase I Double-blinded, Placebo-controlled, Randomized Trial in HIV-uninfected, Healthy Adult Volunteers to Evaluate the Safety and Immunogenicity of an Adjuvanted GSK HIV Vaccine Administered With Ad35-GRIN Investigational Vaccine
Brief Title: Safety and Immunogenicity Study of 2 Investigational Preventive HIV Vaccines
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: International AIDS Vaccine Initiative (Network)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IAVI B002
Record Dates: First submitted 2010-12-20; First posted 2010-12-21 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-02

CONDITIONS: HIV Infections
Keywords: HIV
MeSH Terms: conditions — HIV Infections | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group A (Experimental): Adjuvanted GSK investigational HIV vaccine at Months 0 and 1 followed by Ad35-GRIN investigational HIV vaccine at Month 4.
  Interventions: Biological: Adjuvanted GSK investigational HIV vaccine formulation 1; Biological: Ad35 investigational HIV vaccine; Biological: Placebo (saline)
- Group B (Experimental): Adjuvanted GSK investigational HIV vaccine at Months 0 and 1 followed by Ad35-GRIN investigational HIV vaccine at Month 4.
  Interventions: Biological: Adjuvanted GSK investigational HIV vaccine formulation 2; Biological: Ad35 investigational HIV vaccine; Biological: Placebo (saline)
- Group C (Experimental): Ad35-GRIN investigational HIV vaccine at Month 0 followed by Adjuvanted GSK investigational HIV vaccine at Months 3 and 4.
  Interventions: Biological: Ad35 investigational HIV vaccine; Biological: Adjuvanted GSK investigational HIV vaccine formulation 2; Biological: Placebo (saline)
- Group D (Experimental): Adjuvanted GSK investigational HIV vaccine and Ad35-GRIN investigational HIV vaccine co-administered (simultaneous administration with separate injections)at Months 0, 1, and 4.
  Interventions: Biological: Adjuvanted GSK investigational HIV vaccine formulation 2; Biological: Ad35 investigational HIV vaccine; Biological: Placebo (saline)

INTERVENTIONS:
Biological: Adjuvanted GSK investigational HIV vaccine formulation 1 — Receive at Months 0 and 1
  Arms: Group A
Biological: Adjuvanted GSK investigational HIV vaccine formulation 2 — Receive at Months 0 and 1
  Arms: Group B
Biological: Ad35 investigational HIV vaccine — Receive at Month 0
  Arms: Group C
Biological: Adjuvanted GSK investigational HIV vaccine formulation 2 — Receive at Months 3 and 4
  Arms: Group C
Biological: Adjuvanted GSK investigational HIV vaccine formulation 2 — Receive at Months 0, 1, and 4
  Arms: Group D
Biological: Ad35 investigational HIV vaccine — Receive at Month 4
  Arms: Group A; Group B
Biological: Ad35 investigational HIV vaccine — Receive at Months 0, 1, and 4
  Arms: Group D
Biological: Placebo (saline) — (Vaccine:Placebo=28:7) Groups A, B, C, and D will all have a placebo comparator component (7 volunteers will receive placebo in each group at the specified months.)

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and immunogenicity of an adjuvanted GSK investigational HIV vaccine and Ad35-GRIN in 4 different regimens at months 1, 2, 3, and 4.

DETAILED DESCRIPTION:
Volunteers will be screened up to 42 days before vaccination (up to 90 days for Ad35 neutralizing antibody) and will be followed for 12 months after the last vaccination (16 months total participation).

It is estimated that it will take approximately 5 months to complete enrolment.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females, as assessed by a medical history, physical exam, and laboratory tests
2. At least 18 years of age on the day of screening and has not reached his/her 41st birthday on the day of first vaccination
3. Willing to comply with the requirements of the protocol and available for follow-up for the planned duration of the study (screening plus 16 months)
4. In the opinion of the Principal Investigator or designee and based on Assessment of Informed Consent Understanding results, has understood the information provided and potential risks linked to vaccination and participation in the trial. Written informed consent needs to be provided by the volunteer before any study-related procedures are performed
5. Willing to undergo HIV testing, risk reduction counselling, receive HIV test results and committed to maintaining low risk behaviour for the trial duration
6. If a female of childbearing potential (not menopausal or anatomically sterile), willing to use an effective non-barrier method of contraception (hormonal contraceptive; intra-uterine device), from screening until four months after last vaccination. All female volunteers must be willing to undergo urine pregnancy tests at time points as indicated in the study protocol and must test negative prior to each vaccination.
7. If sexually active male (who is not anatomically sterile), willing to use an effective method of contraception (such as consistent condom use) from the day of first vaccination until 4 months after the last vaccination
8. Willing to forgo donations of blood or any other tissues during the study and, for those who test HIV positive after vaccination, until the anti-HIV antibody titres become undetectable

Exclusion Criteria:

1. Confirmed HIV-1 or HIV-2 infection
2. Any clinically relevant abnormality on history or examination including history of immunodeficiency, malignancy or autoimmune disease; use of systemic corticosteroids (<2 weeks use of topical or inhaled steroids is permitted); immunosuppressive, anticancer, anti-tuberculosis or other medications considered significant by the investigator within the previous 6 months
3. Any clinically significant acute or chronic medical condition that is considered progressive, or in the opinion of the investigator, makes the volunteer unsuitable for participation in the study
4. Detection of Ad35-specific serum neutralizing antibody
5. Reported high-risk behaviour for HIV infection within 6 months prior to first vaccination, as defined by the protocol.
6. If female, pregnant or planning a pregnancy within 4 months after last vaccination; or lactating
7. Unstable asthma (e.g. sudden acute attacks occurring without an obvious trigger) or asthma requiring:

   * Daily steroid or long acting beta-agonist prevention
   * Hospitalization in the last two years
8. Bleeding disorder that was diagnosed by a physician e.g., factor deficiency, coagulopathy or platelet disorder that requires special precautions. (A volunteer who states that he or she has easy bruising or bleeding, but does not have a formal diagnosis and has intramuscular (IM) injections and blood draws without any adverse experience is eligible)
9. History of splenectomy
10. Any abnormal laboratory parameters as defined by the protocol;
11. Receipt of live-attenuated vaccine within the previous 60 days (live attenuated flu vaccine within 14 days) or planned receipt within 60 days after vaccination with Investigational Product; or receipt of other vaccine (e.g. pneumococcal), allergy treatment with antigen injections or tuberculin skin test within the previous 14 days or planned receipt within 14 days after vaccination with Investigational Product
12. Receipt of blood transfusion or blood-derived products within the previous 6 months
13. Participation in another clinical trial of an Investigational Product currently, within the previous 3 months or expected participation during this study
14. Prior receipt of another investigational HIV vaccine candidate (note: receipt of an HIV vaccine placebo will not exclude a volunteer from participation if documentation is available and the IAVI Medical Monitor gives approval)
15. History of severe local or systemic reactogenicity to vaccines (e.g. anaphylaxis, respiratory difficulty, angioedema)
16. History of severe allergic reactions to any substance requiring hospitalization or emergency medical care (e.g. Steven-Johnson syndrome, bronchospasm or hypotension)
17. Known sensitivity to sulphite, aspirin or aminoglycoside antibiotics (e.g. amikacin, arbekacin, gentamicin, kanamycin, neomycin, netilmicin, paromomycin, streptomycin, tobramycin, etc)
18. Confirmed diagnosis of active hepatitis B (HBsAg), hepatitis C (HCV antibodies), active syphilis or active tuberculosis
19. History of severe neurological disorder, seizure or psychiatric disorder (e.g schizophrenia, severe psychosis, bipolar disorder requiring therapy, suicidal attempt or ideation)
20. For those volunteers at clinical centres participating in ophthalmic examinations, any clinically significant abnormality found on baseline ophthalmic examination.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 147 (Actual)
Dates: Start 2011-02; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Safety of an adjuvanted HIV protein vaccine in prime-boost combinations with AD35-GRIN or coadministered with AD35-GRIN | 16 months
  Safety of an adjuvanted (dose escalation for adjvans) HIV protein vaccine given as prime or boost in combination with Ad35-GRIN or co-administered with Ad35-GRIN

SECONDARY OUTCOMES:
Immunogenicity of an adjuvanted HIV protein vaccine given in different prime-boost regimens with Ad35-GRIN or coadminisitered with Ad35-GRIN | 16 months

CONTACTS AND LOCATIONS:
Overall Officials: Gloria S Omosa-Manyonyi, MBChB,DPH,DLSHTM, MSc., Principal Investigator — Kenya AIDS Vaccine Initiative; Juliet Mpendo, MBChB, MPH, Principal Investigator — Uganda Virus Research Institute-IAVI; Eugene Ruzagira, MBChB MPH, Principal Investigator — Medical Research Council-UVRI Uganda Research Unit on AIDS; Elwyn Chomba, BSc, MBChB, DCH, MRCP, Principal Investigator — Zambia-Emory HIV Research Project
Locations (4):
- Kenya AIDS Vaccine Initiative, Nairobi, Kenya
- Uganda (2):
  - Uganda Virus Research Institute-IAVI, Entebbe
  - Medical Research Council, Masaka
- Zambia-Emory HIV Research Project, Lusaka, Zambia

REFERENCES:
- [Derived] Omosa-Manyonyi G, Mpendo J, Ruzagira E, Kilembe W, Chomba E, Roman F, Bourguignon P, Koutsoukos M, Collard A, Voss G, Laufer D, Stevens G, Hayes P, Clark L, Cormier E, Dally L, Barin B, Ackland J, Syvertsen K, Zachariah D, Anas K, Sayeed E, Lombardo A, Gilmour J, Cox J, Fast P, Priddy F. A Phase I Double Blind, Placebo-Controlled, Randomized Study of the Safety and Immunogenicity of an Adjuvanted HIV-1 Gag-Pol-Nef Fusion Protein and Adenovirus 35 Gag-RT-Int-Nef Vaccine in Healthy HIV-Uninfected African Adults. PLoS One. 2015 May 11;10(5):e0125954. doi: 10.1371/journal.pone.0125954. eCollection 2015. PMID 25961283
- See also: International AIDS Vaccine Initiative — http://www.iavi.org